CLINICAL TRIAL: NCT04840966
Title: Simplified Flavor Test for Self-administation in COVID-19 Positive Patients
Brief Title: A Simplified Test to Assess Flavor in COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Paolo Emidio Macchia, Md., Ph.D., Federico II University
Other Study IDs: PM0001/2020
Record Dates: First submitted 2021-04-08; First posted 2021-04-12 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Covid19
Keywords: flavor; smell; flavor test; hyposmia; retro-nasal olfaction
MeSH Terms: conditions — COVID-19; Anosmia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HOS: hospitalized COVID19 patients: Patients positive to COVID19 hospitalized
  Interventions: Diagnostic Test: Flavor test; Other: Self-assesment questionnaire
- HI: Home-isolated COVID19 patients: Home-isolated patients positive to COVID19
  Interventions: Diagnostic Test: Flavor test; Other: Self-assesment questionnaire
- CTRL: Healthy controls: Healthy COVID19 negative subjects
  Interventions: Diagnostic Test: Flavor test

INTERVENTIONS:
Diagnostic Test: Flavor test — A simplified self-administrable flavor test has been proposted to all the enrolled subjects
Other: Self-assesment questionnaire — Questionnaire to score subjective chemosensory function (smell and flavor) before and after COVID-19 using a 0-10 scale with 0 corresponding to "no smell/flavor perception" and 10 corresponding to "excellent smell/flavor perception".
  Groups: HI: Home-isolated COVID19 patients; HOS: hospitalized COVID19 patients

SUMMARY:
The Flavor test has been developed and validated by our group to assess retro-nasal olfactory performances.

The original flavor test has been simplified, with the great advantage to be self-administrable for COVID-19 patients in isolation, without any risk to health professionals.

DETAILED DESCRIPTION:
Smell and taste dysfunctions (STDs) are symptoms associated with COVID-19 syndrome, even if their incidence is still uncertain and variable. In this study, the effects of SARS-CoV-2 infection on chemosensory function have been investigated using both a self-reporting questionnaire on smell and flavor perception, and a simplified flavor test. A total of 111 subjects (19 hospitalized [HOS] and 37 home-isolated [HI] COVID-19 patients, and 55 healthy controls [CTRL]) were enrolled in the study. The flavor test used consists in the self-administration of four solution with a pure olfactory stimulus (coffee), a mixed olfactory-trigeminal stimulus (peppermint), and a complex chemical mixture (banana).

After SARS-CoV-2 infection, HOS and HI patients reported similar frequency of STDs, with a significant reduction of both smell and flavor self-estimated perception.

The aromas of the Flavor test were recognized by HI and HOS COVID-19 patients similarly to CTRL, however the intensity of the perceived aromas was significantly lower in patients compared to controls.

This suggests that a chemosensory impairment is present after SARS-CoV-2 infection, and the modified "flavor test" could be a novel self-administering objective screening test to assess STDs in COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years of age) that gave their written informed consent to the study
* Diagnosis of COVID-19 was confirmed by PCR of nasopharyngeal swab (HI or HOS)
* Negative COVID-19 nasopharyngeal swab (CTRL)
* Subjects with no critical conditions and able to understand the protocol

Exclusion Criteria:

* nasal obstruction or previous nasal diseases

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A total of 111 subjects (19 hospitalized [HOS] and 37 home-isolated [HI] COVID-19 patients, and 55 healthy controls [CTRL]) were enrolled in the study. The mean age for overall population was 41.52±14.45 years.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2020-05-05 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Flavor perception | Apr, 2020- Jan, 2021
  To assess qualitative flavor perception

SECONDARY OUTCOMES:
Flavor perception intensity | Apr, 2020- Jan, 2021
  To assess quantitative flavor perception

OTHER OUTCOMES:
Comparison with self-estimated flavor perception | Apr, 2020- Jan, 2021
  To compare results of the test with self-assessed flavor and smell perception

CONTACTS AND LOCATIONS:
Overall Officials: Paolo E Macchia, M.D., Ph.D., Principal Investigator — Federico II University
Locations (1):
- Dipartimento di Medicina Clinica e Chirurgia, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nettore IC, Cantone E, Palatucci G, Franchini F, Maturi R, Nerilli M, Manzillo E, Foggia M, Maione L, Ungaro P, Colao A, Macchia PE. Quantitative but not qualitative flavor recognition impairments in COVID-19 patients. Ir J Med Sci. 2022 Aug;191(4):1759-1766. doi: 10.1007/s11845-021-02786-x. Epub 2021 Sep 25. PMID 34562193